CLINICAL TRIAL: NCT06822127
Title: Simulation of Facial Soft Tissue in Orthognathic Surgery
Acronym: SPOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-02; 2024-A02357-40 (Other: ANSM)
Record Dates: First submitted 2025-02-11; First posted 2025-02-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: A non-controlled, non-randomised interventional cohort study of patients undergoing planned orthognathic surgery, designed to evaluate the simulation of changes to the soft parts of the face during surgery, using the SPOC simulation model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing orthognathic surgery, (Other): Patients undergoing isolated mandibular or maxillary orthognathic surgery, or maxillo-mandibular surgery with or without genioplasty, whatever the indication (occlusal disorder, sleep apnoea syndrome, functional joint disorder, etc.)
  Interventions: Other: CT scan; Other: VLASTIC test

INTERVENTIONS:
Other: CT scan — 6 months postop CT scan
Other: VLASTIC test — Measurement of the elasticity of the facial integument using the VLASTIC cutometer (Volume-based Light Aspiration device for in vivo Soft Tissue Characterization)

SUMMARY:
Orthognathic surgery consists of rebalancing the position of the jaws, taking into account functional criteria (tooth engagement, tooth/lip ratio, breathing, etc.) and aesthetic criteria. It has become much more accurate in recent years thanks to the advent of osteosynthesis plates and the contribution of three-dimensional imaging. Three-dimensional imaging makes it possible to simulate fairly accurately the surgical procedures and bone displacements required. However, the effect of these bone displacements on the soft tissues (skin, subcutaneous tissue, muscles) does not make it possible, with today's digital tools, to simulate the final aesthetic result and in particular to anticipate the sometimes significant postoperative changes to the face. Many patients are worried about these post-operative morphological changes and would like to have a precise idea of how they will look after surgery. Being able to offer them, before surgery, a visual solution simulating the final aesthetic appearance would be essential in this respect.

The aim of the study is to validate the predictions provided by the digital face model on a series of patients scheduled for orthognathic surgery by comparing the simulation of the morphological result of the operation, provided by our algorithm (SPOC), with the actual result assessed on a scan taken 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 ;
* Patients who have been informed of the study and who have freely given their informed consent to participate in the study;
* Patient undergoing isolated mandibular or maxillary orthognathic surgery, or maxillo-mandibular surgery with or without genioplasty for any indication (occlusal disorder, sleep apnoea syndrome, functional joint disorder, etc.);
* Patient covered by a French social security scheme

Exclusion Criteria:

* Patient with maxillary disjunction ;
* Patients with facial malformations;
* Pregnant or breast-feeding patient;
* Patient under guardianship;
* Patients who do not understand French;
* Patients under court protection
* No pre- or postoperative CT scan or CT scan that cannot be used
* Surgery, trauma, progressive infection or cosmetic injection on the face after orthognathic surgery and before the postoperative scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the predictions provided by the digital face model (SPOC). | 6 months after orthganthic surgery
  Correlation of morphological result simulation of surgery, provided by our algorithm (SPOC), with the actual result assessed on a scan taken 6 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Georges BETTEGA, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (1):
- CH Annecy Genevois, Annecy, France

IPD SHARING:
Plan to Share IPD: No